CLINICAL TRIAL: NCT04901780
Title: Shoulder Stertching
Brief Title: Pragmatic Posterior Capsular Stretch
Acronym: PPCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helping Hand Institute of Rehabilitation Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: rec/hhirs/batch4/002
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2020-12

CONDITIONS: Shoulder Impingement; Shoulder Pain; Adhesive Capsulitis; Rotator Cuff Tears; Posterior Capsule Tear; Glenohumeral Subluxation; Glenohumeral Dysplasia; Acromioclavicular; Sprain (Strain); Internal Rotation Contracture-shoulder; External Rotation Contracture-Shoulder; Flexion Contracture; Extension Contracture-Shoulder
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain; Bursitis; Rotator Cuff Injuries; Shoulder Dislocation; Sprains and Strains

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The enumerator will not know about the interventions used for the side of the body
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPCS (Experimental): Novel intervention
  Interventions: Other: pragmatic posterior capsular stretch
- CBS (Active Comparator): Cross arm stretch gave to individuals
  Interventions: Other: cross body stretch

INTERVENTIONS:
Other: pragmatic posterior capsular stretch — pragmatic posterior stretch is used to increase the length of the posterior capsule
  Arms: PPCS
Other: cross body stretch — crossbody stretch performed by an individual
  Arms: CBS

SUMMARY:
Various stretches are used to lengthen the posterior shoulder capsule. No study has reported the comparison of the pragmatic posterior capsular stretch and cross body stertch

DETAILED DESCRIPTION:
Background: Posterior capsular tightness (PCT) is a problem frequently seen in shoulder disorder. PCT leads to variation in scapular and humeral kinematics. Two techniques considered in our study for regaining normal range of motion at shoulder joint and improving PCT, one is the pragmatic posterior capsular stretch (PPCS) & the other one is cross body stretch (CBS) Objective: The aim of our study id to compare the short term effect of PPCS versus CBS on range of motion on shoulder joint in healthy individuals. And to evaluate the feedback of subjects regarding both the interventions.

Methodology: Through RCT 30 asymptomatic subjects (15 males, 15 females) . A simple random sampling technique was used. Subjects were screen through a functional movement screening tool. The change in hand behind neck and hand behind back will be measured through measuring tape. Shoulder ROM and functional movements for both the stretches will be campared

Results:

ELIGIBILITY:
Inclusion Criteria:

* Age groups of males and females including 20-35 years
* Subjects who fall in grade 1 and 2 of functional movement screening of shoulder during the screening process.

Exclusion Criteria:

* Individual with shoulder pain, fracture or dislocation less than 1 year
* Individuals with any known shoulder pathology
* Subjects receiving current physiotherapy treatment
* Subjects having enough range of motion( can reach T2 hand behind neck)

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
shoulder flexion | 4 week
  range of motion of shoulder flexion
shoulder abduction | 4 week
  range of motion of shoulder abduction
shoulder internal rotation | 4 week
  range of motion of shoulder internal rotation
shoulder external rotation | 4 week
  range of motion of shoulder external rotation
hand behind neck | 4 week
  range of hand behind neck
hand behind back | 4 week
  range of hand behind back

CONTACTS AND LOCATIONS:
Locations (1):
- Helping Hand Institute of Rehabilitation Sciences, Mansehra, Khyber Pakhtoon Khawa, Pakistan

IPD SHARING:
Plan to Share IPD: No